CLINICAL TRIAL: NCT07234968
Title: Randomized Controlled Trial to Evaluate Post-Operative Outcomes of Ureteral Stent vs Ureteral Stent Free Radical Cystectomy
Brief Title: Clinical Trial to Evaluate Post-Operative Outcomes of Ureteral Stent vs Ureteral Stent Free Radical Cystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iRISID-2025-0635; JT 45452 (Other: JeffTrial Number); 2025-117 (Other: PRMC Number)
Record Dates: First submitted 2025-10-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer; Muscle-Invasive Bladder Carcinoma; Urothelial Carcinoma; Pelvic Malignancy; Bladder Transitional Cell Carcinoma; Bladder Neoplasm
Keywords: Bladder; Stent-free Cystectomy; Urinary Tract Infection; Urinary Leak; UTI; Pelvic Malignancy; Bladder Cancer; Urologic Oncology; Muscle-invasive Bladder Cancer; indocyanine green; fluorescence imaging; ureteral stents; RCIC; cystectomy; colorectal; prostate; gynecologic; ileal conduit urinary diversion
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Urinary Tract Infections | interventions — Optical Imaging

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to receive stent or no stent during RCIC. Randomization will be stratified by surgical approach (open vs. robotic vs. hybrid). The randomization schedule will be created by the study statistician using the method of random permuted blocks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1: Ureteral Stent (Experimental): Subjects randomized to the stent arm will receive ureteral stents (double J or single J ureteral catheter, per surgeon preference) during radical cystectomy with ileal conduit urinary diversion (RCIC). Intraoperative use of indocyanine green with fluorescence imaging with be noted. Ureteral stents will be placed intraoperatively and removed at follow up visit per surgeon discretion. Either approach would be considered standard of care for muscle invasive bladder cancer, for which radical cystectomy with urinary diversion is the gold standard of treatment. They will follow the standard of care and be enrolled in the study for 12 months post-op. Risk of post-op complications will be analyzed.
  Interventions: Procedure: Ureteral Stent Placement; Diagnostic Test: Indocyanine Green with Fluorescence Imaging
- Arm 2: No Ureteral Stent (Active Comparator): Subjects randomized to the no-stent arm will undergo radical cystectomy with ileal conduit urinary diversion (RCIC) without placement of ureteral stents. They will follow the standard of care and be enrolled in the study for 12 months post-op. Risk of post-op complications will be analyzed.
  Interventions: Procedure: No Ureteral Stent; Diagnostic Test: Indocyanine Green with Fluorescence Imaging

INTERVENTIONS:
Procedure: Ureteral Stent Placement — Placement of ureteral stents (double J or single J) intraoperatively during radical cystectomy with ileal conduit urinary diversion (RCIC). Stent placement will be a one-time occurrence inserted during RCIC, and be removed typically between 7-21 days post-op at the discretion of the surgeon.
  Other Names: double J; single J; ureteral stents
  Arms: Arm 1: Ureteral Stent
Procedure: No Ureteral Stent — Radical cystectomy with ileal conduit urinary diversion (RCIC) performed without ureteral stent placement.
  Arms: Arm 2: No Ureteral Stent
Diagnostic Test: Indocyanine Green with Fluorescence Imaging — Indocyanine green (ICG) with fluorescence imaging is an advanced technique used to enhance the visualization of the ureters during complex pelvic surgeries, such as those for bladder cancer. The technology helps surgeons identify the ureters, which are the tubes connecting the kidneys to the bladder, and distinguish them from surrounding tissues.
  Other Names: ICG

SUMMARY:
Subjects will be randomized into 2 groups (stent or no stent) prior to radical cystectomy with ileal conduit urinary diversion (RCIC). They will follow the standard of care and be enrolled in the study for 12 months post-op. Risk of post-op complications will be analyzed.

DETAILED DESCRIPTION:
Patients who are indicated for RCIC will be recruited for this prospective RCT. Ureteral stents will be placed intraoperatively and removed at follow-up visit per surgeon discretion. Either approach would be considered standard of care for muscle invasive bladder cancer, for which radical cystectomy with urinary diversion is the gold standard of treatment.

Patients will be randomized 1:1 to receive stent or no stent during RCIC (Stent: N=35, No Stent: N=35). Randomization will be stratified by surgical approach (open vs. robotic vs. hybrid). The randomization schedule will be created by the study statistician using the method of random permuted blocks.

Stent placement, if applicable, will be a one-time occurrence inserted during RCIC, and be removed typically between 7-21 days post-op at the discretion of the surgeon. For this study, subjects will continue to be followed for up to 1-year post-op. Subjects will be enrolled in this study for 12 months.

Post treatment, the patient will have a 2-week follow-up visit (+/- 7 days), 1-month follow-up visit (+/- 7 days), 3-month follow-up visit (+/- 1 week), 6-month follow-up visit (+/- 2 weeks), and 12-month follow-up visit (+/- 2 weeks). Patient will be followed for 12 months post treatment or until their death. Additional visits or follow-ups may be indicated for instances of the need for replacement of ureteral stents and catheters or percutaneous nephrostomies. The need for surgical repair for a ureteral leak or stricture may also occur.

The Principal Investigator hypothesizes that patients with no ureteral stent placement during RCIC will not be associated with a higher risk of post-op complications compared to those with a ureteral stent.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all the following inclusion criteria to be eligible to participate in the study:

  * Provide signed and dated informed consent form
  * Willing to comply with all study procedures and be available for the duration of the study
  * Male or female, age 18 to 85
  * Diagnosed with bladder cancer, other pelvic malignancies necessitating a cystectomy (e.g.: colorectal, prostate, gynecologic) and have elected for a cystectomy with ileal conduit urinary diversion

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  * Current or history of pelvic radiation
  * Retroperitoneal fibrosis
  * Intraoperative surgeon decision based on patient anatomy (unhealthy appearing ureter or compromised vascular supply to ureter or scarring of the ureter)
  * Untreated urinary tract infection (UTI) within 30 days prior to RCIC
  * Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of urinary tract infection (UTI) | 90 days after surgery
  UTI is defined as clinical symptoms consistent with UTI as well as urine culture growing >100K per high powered field bacteria. Subjects who do not complete the 90-day follow-up period but had no evidence of infection at last follow-up will be excluded from the analysis. the Mantel-Haenszel stratified-adjusted estimate of the risk difference for incidence of urinary tract infection (risk in no stent arm - risk in stent arm) will be estimated along with one-sided (upper bound) 80% confidence interval

SECONDARY OUTCOMES:
Incidence of urinary leak | 90 days after surgery
  Measurement will be the presence or absence of a urinary leak. Urinary leak will be identified through clinical symptoms, laboratory abnormalities, or imaging findings. Relevant assessments include vitals, laboratory testing (CBC and BMP/CMP), urinalysis, and imaging reports. Data will be aggregated as the number and percentage of participants with a urinary leak within the time frame.
Incidence of ureteral stricture | 12 months after surgery
  Measurement will be the presence or absence of ureteral stricture. Ureteral stricture will be identified through clinical symptoms, laboratory abnormalities, or imaging findings. Relevant assessments include vitals, laboratory testing (CBC and BMP/CMP), urinalysis, and imaging reports. Data will be aggregated as the number and percentage of participants with ureteral stricture within the time frame.

OTHER OUTCOMES:
Incidence of readmission | within 90 days
  Measurement will be the presence or absence of hospital readmission. Readmission is defined as any unplanned hospital admission during follow-up. Assessments include vitals, adverse event review, labs, urinalysis, and imaging performed at the scheduled post-operative visits. Data will be aggregated as the number and percentage of participants with ureteral stricture within the time frame.
Incidence of secondary intervention or procedure related to UTI or Urine Leak or Ureteral Stricture | within 12 months after surgery
  Measurement will be the presence or absence of secondary intervention or procedure related to UTI or Urine Leak or Ureteral Stricture. These will be identified through hospital readmissions. Readmission is defined as any unplanned hospital admission during follow-up. Assessments include vitals, adverse event review, labs, urinalysis, and imaging performed at the scheduled post-operative visits. Data will be aggregated as the number and percentage of participants with ureteral stricture within the time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Mihir S Shah, MD, Principal Investigator — Thomas Jefferson University

IPD SHARING:
Plan to Share IPD: No